CLINICAL TRIAL: NCT05905627
Title: The Effect of Breathing and Relaxation Exercise on Dyspnea, Fatigue and Self-Care Level
Brief Title: Breathing Relaxation Exercise Heart Failure
Status: Completed | Type: Observational
Sponsor: University of Yalova (Other)
Responsible Party: Principal Investigator, Gürcan Solmaz, PhD, University of Yalova
Other Study IDs: gurcan
Record Dates: First submitted 2023-06-06; First posted 2023-06-15 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Congestive Heart Failure
Keywords: heart failure, breathing exercise, relaxation exercise
MeSH Terms: conditions — Heart Failure | interventions — Exercise; Respiration

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- breathing exercise group: breathing exercise group
  Interventions: Behavioral: exercise
- relaxation exercise group: relaxation exercise group
  Interventions: Behavioral: exercise
- control group: control group

INTERVENTIONS:
Behavioral: exercise — intervention group
  Other Names: breathing and relaxation exercise
  Groups: breathing exercise group; relaxation exercise group

SUMMARY:
The aim of the study is to determine the effect of breathing and relaxation exercises on dyspnea, fatigue and self-care level in heart failure patients.

DETAILED DESCRIPTION:
The Effect of Breathing and Relaxation Exercise on Dyspnea, Fatigue and Self-Care Level in Patients with Heart Failure: A Randomized Controlled Study It was planned according to CONSORT rules as a randomized controlled study to determine its effect on self-care level.

The hypotheses of the research are as follows:

a: Breathing exercise applied to HF patients has an effect on the mean dyspnea score. b: Breathing exercise applied to HF patients has an effect on the mean fatigue score. c: Breathing exercise applied to HF patients has an effect on self-care mean scores. d: Relaxation exercise applied to HF patients has an effect on the mean dyspnea score. e: Relaxation exercise applied to HF patients has an effect on the mean fatigue score.

f: Relaxation exercise applied to HF patients has an effect on self-care mean scores.

ELIGIBILITY:
Inclusion Criteria:

(a) 18 years of age or older; (b) Patients with HF stage NYHA II-III; (c) hospitalized for two weeks; (d) Not pregnant; (e) Not applying any integrated treatment; (f) Patients who have been taking the same heart failure medication for at least three months.

Exclusion Criteria:

The exclusion criteria of patients are as follows: (a) Not expected to participate in a breathing or progressive relaxation exercise study in expert opinion; (b) Patients with COPD, (d) Patients with severe mental disorders.

Individuals' eligibility for inclusion and exclusion criteria will be evaluated through patient file records and interviews with the physician.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The universe of the research; all heart failure patients. In order to determine the sample of the study, a similar study Lopes et al. (2018) considering the data obtained from the study, power=0.80, α=0.05 and β=0.20 were calculated. It was determined that 80% power could be reached if the study was conducted with at least 20 individuals in each group, at a significance level of p<0.05, with a medium effect size (ES: 0.5) in independent groups, with a 95% confidence interval. As a result of the calculation, taking into account the problems that may arise during the study process, it is planned to sample a total of 75 patients, 25 patients in each group (intervention group (yoga breathing and progressive relaxation exercise group) and control group).
Sampling Method: Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2023-06-06 (Actual); Primary Completion 2023-06-11 (Actual); Study Completion 2023-06-21 (Actual)

PRIMARY OUTCOMES:
The effect of ephesus exercise on the mean fatigue score | 3 months
  The effect of ephesus exercise on the mean fatigue score

CONTACTS AND LOCATIONS:
Locations (1):
- Yalova University, Yalova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It is planned to collect data between May and July 2023. Initially, patients' compliance with the inclusion and exclusion criteria will be determined through patient file records and interviews with the physician, and randomization will be performed. The research will be carried out in the hospital with the patients whose sample group is determined. In the first interview at the hospital, BPF, Borg Dyspnea Scale, Piper Fatigue and Self-Care Scale will be evaluated by the researcher through face-to-face interviews with the patients.